CLINICAL TRIAL: NCT00750191
Title: A Randomized, Placebo-controlled Trial of Transdiscal Radiofrequency Annuloplasty for Treatment of Discogenic Lower Back Pain
Brief Title: Placebo-controlled Trial of Transdiscal Radiofrequency Annuloplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylis Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 07-594; IRB 07-594
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2013-11

CONDITIONS: Lower Back Pain
Keywords: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intradiscal Biacuplasty (Active Comparator): On the day of the procedure, patients were given midazolam for relaxation and, if needed, fentanyl IV during the procedure. For treatment subjects, two TransDiscal probes were positioned under fluoroscopic guidance in the posterior annulus of the intervertebral disc. The probes were attached to the Radiofrequency generator and Radiofrequency energy was delivered. Placement of the probes within the disc annulus was confirmed using oblique, lateral, and anterior-posterior fluoroscopic images.
  Following completion of procedure the patient was transferred to recovery and monitored for 45 minutes then discharged home with instructions. It was expected that the patient limit their activities during the first week after the procedure.
  Interventions: Device: The Transdiscal Radiofrequency Annuloplasty
- Sham (Placebo Comparator): Sham procedures mimicked active treatment procedures, except that the probes were positioned just outside of the disc and no radiofrequency energy was delivered through the electrodes. Thus, sham patients were provided similar tactile, auditory and visual experiences as treatment patients, without receiving the active RF treatment.
  Following completion of procedure the patient was transferred to recovery and monitored for 45 minutes then discharged home with instructions. It was expected that the patient limit their activities during the first week after the procedure.
  The study will be unblinded at 6 months. If the patients in the IDB group show significant improvement compared to placebo they will be offered IDB.
  Interventions: Device: The Transdiscal Radiofrequency Annuloplasty

INTERVENTIONS:
Device: The Transdiscal Radiofrequency Annuloplasty — Adjustment in dosage form, frequency and or duration.
  Other Names: Intradiscal Biacuplasty Active Comparator
  Arms: Intradiscal Biacuplasty
Device: The Transdiscal Radiofrequency Annuloplasty — interventions include adjustment to dosage form,frequency,duration or switching to treatment arm A
  Other Names: Sham: Placebo Comparator
  Arms: Sham

SUMMARY:
Each patient was assigned to one of the two groups: IDB or Sham. On the day of the procedure, an IV was inserted in pre-procedural area and patient transported to the procedure room. The procedure will be completed under fluoroscopy in prone position. Patients were given 1-4 mg of midazolam for relaxation before the procedure and, if needed, 50-100 mcg of fentanyl IV during the procedure. The patients was randomly assigned to treatment or placebo using computer-generated codes maintained in sequentially numbered opaque envelopes. The physician performing procedure was informed of the assignment. In IDB group, guided by the fluoroscopic imaging, two transdiscal probes was positioned in the posterior annulus using a posterolateral, oblique approach. First, two electrically insulated 17G transdiscal introducers was used to gain an access to the disc space. Than, two radiofrequency probes will be positioned through each of the introducers bilaterally to create a bipolar configuration. Placement of the transdiscal probes within the disc annulus will be confirmed using oblique, lateral, and anterior-posterior fluoroscopic images. Sham group had their introducers and electrodes positioned just outside of the disc. This was also be documented using fluoroscopy. Investigator attached the electrodes to inactive heater control device that provide a similar auditory and visual experience for the patient. Patients were therefore remain blinded to actual treatment and physician performing procedure was not involved in patient's follow-up. Patients were awake and communicating with the physician conducting the procedure and if pain in legs were present and increased during the procedure, the heating protocol would be stopped. Following completion of procedure the patient was transferred to recovery and monitored for 45 minutes, then discharged home with instructions. The patients were followed over a period of 12 months.

DETAILED DESCRIPTION:
Back Pain

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be as follows:

  * Age 18 + years
  * History of chronic low back pain unresponsive to nonoperative care (including physical therapy and anti-inflammatory medication) for longer than 6 months of at least 5 on VAS
  * No surgical interventions within the last 3 months
  * Back pain more than leg pain which is commonly exacerbated by sitting
  * Pain reproduction present on provocative discography in degenerated disc but not in control discs
  * Disc height at least 50% of adjacent control disc
  * Evidence of single level degenerative disc disease or two level disease without evidence of additional degenerative changes in other disc spaces on MRI

Exclusion Criteria:

* The exclusion criteria are :

  * Evidence of compressive radiculopathy with predominant leg pain
  * Nucleus pulposus herniation on the MRI
  * Disc bulges > 5 mm
  * Prior lumbar surgery of any kind
  * Presence of concordant cervical or thoracic pain
  * Symptoms or signs of the lumbar canal stenosis
  * Evidence of structural abnormality at the symptomatic level like spondylolisthesis
  * Chronic severe conditions such as rheumatoid arthritis and fibromyalgia
  * Patients with pending workers compensation claim, litigation or disability income remuneration
  * Psychological issues by exam or history
  * Beck Depression Inventory (BDI) >20
  * Pregnancy
  * Systemic infection or localized infection at the anticipated entry needle site
  * Allergies to contrast media or to any medication to be used in the procedure
  * Traumatic spinal fracture
  * History of coagulopathy, unexplained bleeding
  * Progressive neurological deficits
  * History of opioid abuse
  * Presence of free disc fragments on MRI
  * More than 2 discs degenerated on MRI
  * Immunosuppression (eg. AIDS, cancer, diabetes, other surgery within last 3 months)
  * Smoking
  * BMI (body mass index) >30 kg/m2
  * Subject unwilling to consent to the study
  * Participation in another investigation within 30 days of signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Kapural, MD, Principal Investigator — Center for Clinical Research; Bruce Vrooman, M.D., Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic Pain Management, Cleveland, Ohio

REFERENCES:
- [Derived] Kapural L, Vrooman B, Sarwar S, Krizanac-Bengez L, Rauck R, Gilmore C, North J, Girgis G, Mekhail N. A randomized, placebo-controlled trial of transdiscal radiofrequency, biacuplasty for treatment of discogenic lower back pain. Pain Med. 2013 Mar;14(3):362-73. doi: 10.1111/pme.12023. Epub 2012 Dec 28. PMID 23279658

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 32 treatment subjects, 4 were removed from the study due to violation of eligibility criteria and 1 removed for withdrawing patient consent. Among the 32 sham subjects, 2 patients were removed from the study due to violation of eligibility criteria.
Groups:
- Intradiscal Biacuplasty: Two electrodes, located at the ends of two thin probes, are placed on both sides of the posterior annulus fibrosus of the intervertebral disc by inserting them through the skin to the intervertebral disc under x-ray guidance. Radiofrequency (RF) current flows in the disc between the two electrodes, heating the tissue in the disc to the desired temperature.
  After the procedure, you will be asked to rest until the anesthesia wears off and then re-assessed for pain. Once you are awake and communicating with the physician conducting the procedure. Following completion of procedure you will be transferred to recovery and monitored for 45 minutes then discharged home with instructions. It is expected that you will limit your activities during the first week after the procedure.
- Sham: The same procedures will be followed as Group A (see above) except you will receive placebo (no treatment at all) during procedure.
  The study will be unblinded at 6 months. If the patients in the IDB group show significant improvement compared to placebo they will be offered IDB.
Period: Overall Study
Arm/Group | Intradiscal Biacuplasty | Sham
Started | 27 | 30
Completed | 22 | 20
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intradiscal Biacuplasty | Sham | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 30 | 57
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10) | 39 (10) | 39 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: Physical Function
Description: Physical function as measured by the Short Form (36) Health Survey questionnaire physical function component.
  Scale range for physical function component: 0 (minimum: worse outcome) to 100 (maximum: best outcome).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal Biacuplasty | Sham
Number analyzed (Participants) | 27 | 30
units on a scale | 62.04 (21.89) | 48.67 (22.97)

2. Secondary Outcome: Pain
Description: Pain level as measured by the Numerical Rating Scale. Scale range: 0 (minimum: best outcome) to 10 (maximum: worse outcome)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal Biacuplasty | Sham
Number analyzed (Participants) | 27 | 30
units on a scale | 4.94 (2.15) | 6.58 (2.11)

3. Secondary Outcome: Disability
Description: Disability as measured by the Oswestry Disability Index. Scale range: 0 (minimum: best outcome) to 100 (maximum: worst outcome)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal Biacuplasty | Sham
Number analyzed (Participants) | 27 | 30
units on a scale | 32.94 (16.14) | 41.17 (13.94)

4. Other Pre Specified Outcome: Opioid Usage
Description: Patient reported Opioid usage (converted to morphine equivalents)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intradiscal Biacuplasty | Sham
Number analyzed (Participants) | 27 | 30
mg | 36.87 (40.56) | 49.48 (91.70)

ADVERSE EVENTS:
Arm/Group | Intradiscal Biacuplasty | Sham
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 0/27 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less